CLINICAL TRIAL: NCT02447016
Title: Decrease of Neuropsychiatric and Neurocognitive Side Effects Prevalence
Brief Title: Decrease of Neuropsychiatric Side Effects After Switching From Atripla to Eviplera
Acronym: DeepSwitch
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no more participants taking atripla
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Itsik Levi Dr, Head HIV/STDs unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-1462-IL-SMC
Record Dates: First submitted 2015-05-10; First posted 2015-05-18 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: HIV
MeSH Terms: interventions — Tenofovir; Emtricitabine, Rilpivirine, Tenofovir Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eviplera (complera) (Experimental): Tab eviplera QD
  Interventions: Drug: Tenofovir disoproxil/emtricitabine/rilpivirine
- atripla (Active Comparator): Tab Atripla QD
  Interventions: Drug: Tenofovir disoproxil/emtricitabine/efavirenz

INTERVENTIONS:
Drug: Tenofovir disoproxil/emtricitabine/rilpivirine
  Other Names: eviplera, complera
  Arms: eviplera (complera)
Drug: Tenofovir disoproxil/emtricitabine/efavirenz
  Other Names: Atripla
  Arms: atripla

SUMMARY:
The aim of this prospective, open label study is to check for differences in neuropsychiatric and neurocognitive measurements among patients that will be switched from Atripla to Eviplera among 40 patients.

DETAILED DESCRIPTION:
40 patients on Atripla for at least 12 weeks with undetectable HIV-1 viral load will be randomly assigned to one of two groups in a ratio of 1:1: half of the patients will be switched to Eviplera and half will remain on Atripla. Neuropsychiatric symptoms will be evaluated using specific questionnaires (anxiety and depression scales, sleeping quality scale, etc) and neurocognitive functions will be assessed using standard tests (Trail A and B, memory tests, etc). Patient satisfaction will be assessed using a visual analog scale. Treatment efficacy will be evaluated by measuring the rate of patients with HIV vilral load under 50 copies/mL.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Receiving Atripla continuously for >12 weeks preceding the screening visit
* Plasma HIV-1 RNA levels (at least in two measurements) <50 copies/mL for >8 weeks prior to the screening visit and at the screening visit
* Atripla or Truvada + Efavirenz was the first antiretroviral regimen and no HIV-1 RNA > 50 copies/mL measured at two consecutive time points after first achieving HIV RNA <50 copies/mL
* Had a genotype prior to starting study drugs and no known resistance to any of the study drugs
* Normal ECG
* Hepatic transaminase (AST and ALT) <5 X upper limit of normal (ULN)
* Total bilirubin <1.5 mg/dL
* eGFR > 60 mL/min
* Neutrophil count > 1000/mm3, platelets >50,000/mm3. Haemoglobin > 8.5 g/dL
* Age > 18
* Males and Females of childbearing potential must have agreed to utilize highly effective contraception methods (two separate forms of contraception, one of which must be an effective barrier method, or be nonheterosexually active, practice sexual abstinence, or have a vasectomized partner) from screening throughout the duration of the study period and for 60 days following the last dose of study drug.

Exclusion Criteria:

* Subjects with known allergy to one of the study drugs
* AIDS defining event diagnosed within 21 days prior to screening
* Females who are pregnant or breast feeding
* Acute hepatitis diagnosed within 21 days prior to screening
* Subjects receiving drug treatment for HCV or subjects anticipated to receive treatment for HCV during the course of the study
* Implanted defibrillator or pacemaker
* Current alcohol or drug abuse judged by the investigator to potentially interfere with subject adherence
* Participation in another interventional trial
* Ongoing therapy or anticipated need to initiate drugs during the study that are contraindicated or not recommended for use with study drugs (Carbamazepine, Dexamethasone, Esomeprazole, Fosphenytoin, Lansoprazole, Omeprazole, Oxcarbazepine, Pantoprazole, Phenobarbital, Phenytoin, Piperaquine, Primnidone, Rabeprazole, Rifabutin, Rifampin, Rifapentine, St John's Wort
* Any Severe Psychiatric disease that judged by the investigator to potentially interfere with subject adherence to protocol or to drugs or that may interfere with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
depression (questionaire) | 12 month
  PHQ which is a validated questionaire for depression
anxiety (questionaire) | 12 month
  STAI which is a validated questionaire for anxiety
sleeping quality (questionaire) | 12 month
  a validated questionaire

SECONDARY OUTCOMES:
Hopkins Verbal Learning Test - Revised (test result in numbers) | 12 month
  a validated test for memory testing
Satisfaction (scale) | 12 month
  Visual Analogue Scale (VAS)
viral load (copies/mL) | 24 month
  efficacy of treatment in keeping undetectable viral load
color trail test - 2 parts (test result in numbers) | 12 month
  a line drawing test which connects points in a certain order. It serves as a general neurocognitive function test
grooved pegboard test (test result in numbers) | 12 month
  a specific test which serves as a general neurocognitive function test and was validated in HIV patients
clock drawing test (test result in numbers) | 12 month
  a general test for dementia
CD4 cell count (number of cells per mm3) | 12 month
  efficacy of treatment in keeping CD4 count from falling after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel